CLINICAL TRIAL: NCT01642680
Title: Optimal Timing of a Tailored Physical Activity Program During Chemotherapeutic Cancer Treatment to Reduce Long-term Cardiovascular Morbidity
Brief Title: Optimal Timing of Physical Activity in Cancer Treatment
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012-0010; 41087 (Registry Identifier: ABR)
Record Dates: First submitted 2012-07-04; First posted 2012-07-17 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Syndrome; Vascular Disorders; Cardiovascular Risk Factors; Fatigue
Keywords: Physical activity program; Chemotherapy; Metabolic syndrome; Reducing cardiovascular risk factors; low physical activity level
MeSH Terms: conditions — Metabolic Syndrome; Vascular Diseases; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity during chemotherapy (Experimental): This group will start with a physical activity program 3 months before the end of their chemotherapeutic regimen. After chemotherapy they will continue the PA program for another 3 months.
  Interventions: Other: A tailored physical activity program during chemotherapy
- Physical activity after chemotherapy (Active Comparator): This group will start with a physical activity program after the end of their chemotherapeutic regimen. The physical activity program wil take 6 months to complete.
  Interventions: Other: A tailored physical activity program after chemotherapy

INTERVENTIONS:
Other: A tailored physical activity program during chemotherapy — The early group will start the PA program during chemotherapy for 3 months, and after completion of chemotherapy for 3 months (total 6 months). The PA program will consist of two components: improvement of physical fitness and empowerment to adopt a healthy lifestyle. Longitudinal effects of this PA program will be evaluated at 5 time points: before chemotherapy; at start of the PA program and at 3, 6 and 18 months after start of the PA program. Safety parameters will be monitored throughout the study period.
  Arms: Physical activity during chemotherapy
Other: A tailored physical activity program after chemotherapy — The late group will start the PA program after completion of the chemotherapy for 6 months. The PA program will consist of two components: improvement of physical fitness and empowerment to adopt a healthy lifestyle. Longitudinal effects of this PA program will be evaluated at 5 time points: before chemotherapy; at start of the PA program and at 3, 6 and 18 months after start of the PA program. Safety parameters will be monitored throughout the study period.
  Arms: Physical activity after chemotherapy

SUMMARY:
The number of long-term cancer survivors is growing. As a result, treatment-related morbidity - such as cardiovascular disease, metabolic syndrome, functional decline and fatigue - is impacting quality of life and impairing survival. Metabolic syndrome in the general population is currently treated with lifestyle advice to increase physical activity (PA) and reduce caloric intake. This approach is still underused as standard care for cancer survivors. The aim of this study is investigate whether a tailored PA program that starts early (during curative chemotherapy with cardiovascular toxic potential) is superior in terms of reducing long-term cancer-treatment-related metabolic syndrome and cardiovascular morbidity to a program that starts late (after completion of chemotherapy).

DETAILED DESCRIPTION:
Improved treatment is partly responsible for the increased survival and life expectancy in cancer patients. However, such treatment can be harmful as well, and cancer survivors therefore, face an increased risk of second malignancies and other chronic diseases, e.g. cardiovascular diseases and metabolic syndrome.

Due to the growing number of cancer patients and survivors, attention for rehabilitation, especially physical training, is growing. Several meta-analyses show the beneficial effects of physical training on several outcomes such as physical fitness, muscle strength, fatigue and quality of life, and a few studies showed the effect of exercise on physical active behaviour. However, studies on the effect of timing of exercise are lacking.

The present study aims to insert a tailored physical activity program early versus late in the chemotherapy based cancer treatment and will yield data about its safety and efficacy. We hypothesize that a tailored physical activity program during early cancer treatment may more be effective to reduce long-term cancer treatment toxicities and morbidity in cancer survivors compared to a program after cancer treatment.

Primary Objective: To investigate whether a tailored physical activity program that starts during chemotherapy (early) is superior in terms of physical fitness, as determined by VO2 peak at one year, to a program that starts after completion of chemotherapy (late).

Secondary Objectives: To examine the effect of the physical activity program on muscle strength and activity level, change in metabolic and cardiovascular damage parameters, cardiovascular risk factors and quality of life including self-efficacy, motivation for exercise, and fatigue.

Design: This protocol describes a multicenter, randomized study with 2 arms. Patients who will be treated with curative systemic chemotherapeutic treatment for testicular cancer, early colon cancer, early breast cancer or B-NHL will be randomized into an early or late PA program group. The early group will start the PA program during chemotherapy (for 12 weeks) until 12 weeks after completion of chemotherapy (total 24 weeks of training). The late group will start the same program (total of 12 weeks) after completion of chemotherapy. The longitudinal effects of the physical activity (PA) program for all participants will be evaluated at different time points in the UMCG: before start of chemotherapeutic treatment; at the start of the PA program and at 3, 6, 18 months after starting the PA program and 18 months after the last chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with testicular, early colon, breast cancer or B-NHL with an indication for systemic chemotherapy with a curative intent
* Normal blood count at start of systemic treatment
* Patients need to have an adequate physical health, which is defined by diastolic blood pressure >45 mm Hg or <95 mm Hg; heart frequency in at rest < 100 per minute; body temperature below 38°C; respiration frequency in rest below 20 per minute
* Adequate cardiac function with a LVEF above the lower limit of normal
* Written informed consent

Exclusion Criteria:

* Infections requiring actual antibiotics
* Signs of ongoing bleeding or fresh petechiae; unexplained bruises
* Critical organ impairment due to their malignancy
* Not recovered from earlier surgical intervention
* Non adequate control of any symptoms of the malignancy
* Inability to travel independently to the rehabilitation centre
* Cognitive disorder or emotional instability that might impede the participation in the training program
* Recent cardiovascular event

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Difference in VO2 peak between the groups after completion of the PA program, measured by cardiopulmonary exercise testing (CPET). | 1,5 year
  The aim of this study is investigate whether a tailored PA program that starts early (during curative chemotherapy with cardiovascular toxic potential) is superior in terms of reducing long-term cancer-treatment-related metabolic syndrome and cardiovascular morbidity to a program that starts late (after completion of chemotherapy).
  The VO2 at the peak of the exercise will be defined as peak oxygen uptake (VO2 peak), measured by cardiopulmonary exercise testing (CPET) on a stationary bicycle ergometer. The CPET is considered to be the most precise measure of cardio-respiratory fitness and is recommended for use in order to determine a patient's objective or subjective difference in exercise capacity

SECONDARY OUTCOMES:
Muscle strength using a hand-held dynamometer | 1,5 year
  Maximal voluntary isometric muscle force of the right and left extremity of extension of the knee, flexion of the knee, flexion of the elbow and extension of the elbow will be measured using a hand-held dynamometer. The "break method" will be used for all measurements. To employ this technique, the examiner gradually overcomes the force exerted by the patient until the extremity gives way. All measurements will be performed at least three times, with recovery intervals of at least 10 seconds. The peak forces (in Newtons) will be recorded and mean values of three technically correct measurements will be taken for analysis.
Intima media thickness will be measured with vascular ultrasound | 1,5 year
  Vascular damage will be determined with the intima-media thickness (IMT) of the common carotid artery and femoral artery, performed with an Ultrasound technique.
Cholesterol levels, measured in blood | 1,5 year
  Measured in blood, in mmol/L
Triglyceride levels, measured in blood | 1,5 year
  Measured in blood, in mmol/L
Glucose levels, measured in blood | 1,5 year
  Measured in blood, in mmol/L
Body mass index, calculated with formula (see below) | 1,5 year
  BMI (body mass index): weight in kilograms divided by height in meters squared
Health related quality of life measured with the EORTC QLQ-C30 | 1,5 year
  Quality of life will be measured with the European Organization for Research and Treatment of Cancer (EORTC), Quality of Life Questionnaire Core 30 (QLQ-C30) version 3.0 questionnaire
Patient reported self-efficacy measured using the ALCOS instrument | 1 year
  Patient reported general self-efficacy, measuring the patients' expectations of their general capacities, will be evaluated using the Dutch version of the General Self-Efficacy Scale (GSES), the "Algemene Competentie Schaal" (ALCOS)
Patient reported fatigue measured with the Multi-dimensional Fatigue Inventory | 1,5 year
  The Multi-dimensional Fatigue Inventory is a validated 20-item questionnaire on different domains of fatigue
Patient reported physical activity level with the PASE questionnaire | 1,5 year
  Physical activity will be assessed with the Sum score of the Physical Activity Scale for the Elderly questionnaire (PASE). This questionnaire consists of questions on leisure time, household and work-related activities.
DNA collection | 1,5 year
  Whole blood will be drawn of patients and collected in EDTA tubes. DNA isolations and the Global Screening Array will be performed at the Human Genomics Facility (HuGeF) of the Genetic Laboratory of the Department of Internal Medicine at Erasmus MC, Rotterdam, the Netherlands
Diffusion capacity of the lungs | 1,5 year
  Corrected for hemoglobin.
Forced vital capacity (FVC) will be assessed by use of dynamic spirometry | 1,5 year
  Measured by means of dynamic spirometry
Forced expiratory volume in one second (FEV1) will be assessed by use of dynamic spirometry, | 1,5 year
  Measured by means of dynamic spirometry
FEV1/FVC ratio will be assessed by use of dynamic spirometry, | 1,5 year
  Measured by means of dynamic spirometry
Senescence with markers of the senescence- associated secretory phenotype | 1,5 year
  Senescence will be measured in a subset of testicular cancer patients.
  Markers of scenescence will be obtained from a skin biopsy and fat biopsy. Also, additional blood samples will be assessed to establish markers of the senescence- associated secretory phenotype.
Cardiac function with echocardiography (Ultrasound technique) | 1,5 year
  Cardiac function will be measured at baseline and at the final measurement (e.g. left ventricular ejection fraction)
Body composition will be assessed with a DEXA scan | 1,5 year
  With the DEXA scan, measurements of body composition will be obtained.
PAI-antigen, measured in blood serum | 1,5 year
  Endothelial activation will be determined with PAI antigen in blood serum, in ug/L
t-PA, measured in blood serum | 1,5 year
  Endothelial activation will be determined with t-PA antigen in blood serum, in ug/L
Factor VIII, measured in blood serum | 1,5 year
  Endothelial activation will be determined with factor VIII in blood serum, in %
Von Willebrand factor, measured in blood serum | 1,5 year
  Endothelial activation will be determined with von Willebrand facor in blood serum, in %
Fibrinogen, measured in blood serum | 1,5 year
  Endothelial activation will be determined with fibrinogen in blood serum, in g/L
Advanced glycation end products (AGEs) will be determined by measuring skin auto fluorescence. | 1,5 year
  Advanced glycation end products will be measured with an AGEreader
Blood pressure, measured with a blood pressure cuff | 1,5 years
  Systolic and diastolic blood pressure in mmHg
Fat percentage with skinfold measurement | 1.5 years
  Skinfold measurement of biceps, triceps, sub scapula and supra iliaca

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Walenkamp, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] van der Schoot GGF, Ormel HL, Westerink NL, Wempe JB, Lefrandt JD, May AM, Vrieling AH, Meijer C, Gietema JA, Walenkamp AME. Physical exercise in patients with testicular cancer treated with bleomycin, etoposide and cisplatin chemotherapy: pulmonary and vascular endothelial function-an exploratory analysis. J Cancer Res Clin Oncol. 2023 Dec;149(19):17467-17478. doi: 10.1007/s00432-023-05469-5. Epub 2023 Oct 27. PMID 37889308
- [Derived] van der Schoot GGF, Ormel HL, Westerink NL, May AM, Elias SG, Hummel YM, Lefrandt JD, van der Meer P, van Melle JP, Poppema BJ, Stel JMA, van der Velden AWG, Vrieling AH, Wempe JB, Ten Wolde MG, Nijland M, de Vries EGE, Gietema JA, Walenkamp AME. Optimal Timing of a Physical Exercise Intervention to Improve Cardiorespiratory Fitness: During or After Chemotherapy. JACC CardioOncol. 2022 Oct 18;4(4):491-503. doi: 10.1016/j.jaccao.2022.07.006. eCollection 2022 Nov. PMID 36444224